CLINICAL TRIAL: NCT04134260
Title: Randomized Phase III Trial Incorporating Apalutamide and Advanced Imaging Into Salvage Treatment for Patients With Node-Positive Prostate Cancer After Radical Prostatectomy (INNOVATE*) *INtensifying Treatment for NOde Positive Prostate Cancer by VArying the Hormonal ThErapy
Brief Title: Testing the Addition of the Drug Apalutamide to the Usual Hormone Therapy and Radiation Therapy After Surgery for Prostate Cancer, INNOVATE Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU008; NCI-2019-06838 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU008 (Other: NRG Oncology); NRG-GU008 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Specimen Handling; Steroids; Hormones; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (hormone therapy, radiation therapy) (Active Comparator): Patients receive standard of care hormone therapy per physician discretion for 24 months. Patients also undergo standard of care pelvis and prostate bed radiation therapy 5 days per week over 5-6 or 7-8 weeks beginning within 90 days of randomization in the absence of disease progression or unacceptable toxicity. Patients in both arms may undergo CT, MRI, bone scan, and PET as clinically indicated throughout the study. Patients may also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Hormone Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Arm II (hormone therapy, radiation therapy, apalutamide) (Experimental): Patients undergo standard of care hormone therapy and radiation therapy as in Arm I. Patients also receive apalutamide PO QD on days 1-90 of each cycle. Cycles repeat every 90 days for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients in both arms may undergo CT, MRI, bone scan, and PET as clinically indicated throughout the study. Patients may also undergo blood sample collection throughout the study.
  Interventions: Drug: Apalutamide; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Hormone Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
  Arms: Arm II (hormone therapy, radiation therapy, apalutamide)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Hormone Therapy — Receive hormone therapy
  Other Names: Chemotherapy-Hormones/Steroids; Endocrine Therapy; Hormonal; Hormonal Therapy; hormone treatment; Hormones
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo pelvis and prostate bed radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase III trial studies whether adding apalutamide to the usual treatment improves outcome in patients with lymph node positive prostate cancer after surgery. Radiation therapy uses high energy x-ray to kill tumor cells and shrink tumors. Androgens, or male sex hormones, can cause the growth of prostate cancer cells. Drugs, such as apalutamide, may help stop or reduce the growth of prostate cancer cell growth by blocking the attachment of androgen to its receptors on cancer cells, a mechanism similar to stopping the entrance of a key into its lock. Adding apalutamide to the usual hormone therapy and radiation therapy after surgery may stabilize prostate cancer and prevent it from spreading and extend time without disease spreading compared to the usual approach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare metastasis-free survival (MFS) of salvage radiation therapy (RT) and gonadotropin releasing hormone (GnRH) agonist/antagonist versus (vs.) RT/GnRH agonist/antagonist with apalutamide for patients with pathologic node-positive prostate cancer after radical prostatectomy with detectable prostate-specific antigen (PSA).

SECONDARY OBJECTIVES:

I. Compare health-related quality of life (Expanded Prostate Cancer Index Composite [EPIC]-26, EuroQol [EQ]-5 Dimension [D]-5 Level [L], Brief Pain Inventory, Patient Reported Outcome Measurement Information System [PROMIS]-Fatigue) among the treatment arms.

II. Compare overall survival, biochemical progression-free survival, time to local-regional progression, time to castrate resistance, and cancer-specific survival among the treatment arms.

III. Compare the short-term and long-term treatment-related adverse events among the treatment arms.

EXPLORATORY OBJECTIVES:

I. Validate Decipher score for an exclusively node-positive population and use additional genomic information from Affymetrix Human Exon 1.0st array to develop and validate novel prognostic and predictive biomarkers.

II. Validate the PAM50-based classification of prostate cancer into luminal A, luminal B, and basal subtypes as prognostic markers and determine whether the luminal B subtype is a predictive marker for having a larger improvement in outcome from the addition of apalutamide.

III. To optimize quality assurance methodologies and processes for radiotherapy and imaging with machine learning strategies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care hormone therapy per physician discretion for 24 months. Patients also undergo standard of care pelvis and prostate bed radiation therapy 5 days per week over 5-6 or 7-8 weeks beginning within 90 days of randomization in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo standard of care hormone therapy and radiation therapy as in Arm I. Patients also receive apalutamide orally (PO) once daily (QD) on days 1-90 of each cycle. Cycles repeat every 90 days for 8 cycles in the absence of disease progression or unacceptable toxicity.

Patients in both arms may undergo computed tomography (CT), magnetic resonance imaging (MRI), bone scan, and positron emission tomography (PET) as clinically indicated throughout the study. Patients may also undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 6 months for 3 years, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically) proven diagnosis of prostate adenocarcinoma. Any type of radical prostatectomy is permitted, including retropubic, perineal, laparoscopic or robotically assisted
* Any T-stage is eligible (American Joint Committee on Cancer [AJCC] 8th edition [ed])
* Appropriate stage for study entry based on fluciclovine F-18 PET scan (FACBC, Axumin) F-18 prostate-specific membrane antigen (PSMA) PET (PyLarify) scan, Gallium-68 PSMA PET scan, flotufolastat F-18 PSMA PET scan (Posluma), or C-11 or F-18 Choline PET within 90 days prior to registration that is negative for distant metastatic (M1a, M1b, M1c) disease. For patients with PSA < 0.20 ng/mL at time of registration, PET scan is recommended but not required
* Pathologically node positive disease with nodal involvement only in the pelvis in the prostatectomy specimen or nodal disease on imaging at time of recurrence (including external iliacs, internal iliacs, and/or obturator nodes); peri-prostatic and peri-rectal nodes can also be considered regional lymphadenopathy and are allowed
* History/physical examination within 90 days prior to registration
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 within 90 days prior to registration
* Detectable PSA after radical prostatectomy. Detectable PSA is defined as serum PSA > 0 ng/mL at least 30 days after prostatectomy
* Patients who have already started on post-prostatectomy GnRH agonist/antagonist for =< 180 days prior to registration are eligible (Note: patients who started on an oral antiandrogen are eligible if started =< 180 days and stopped prior to registration)
* Hemoglobin >= 9.0 g/dL, independent of transfusion and/or growth factors (within 90 days prior to registration)
* Platelet count >= 100,000 x 10^9/uL independent of transfusion and/or growth factors (within 90 days prior to registration)
* Serum potassium >= 3.5 mmol/L within 90 days prior to registration
* Creatinine clearance (CrCl) >= 30 mL/min estimated by Cockcroft-Gault (please use actual weight for calculation unless greater than 30% above ideal body weight then use the adjusted body weight) (within 90 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (Note: In subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject is eligible) (within 90 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (within 90 days prior to registration)
* Serum albumin >= 3.0 g/dL (within 90 days prior to registration)
* Discontinue or substitute concomitant medications known to lower the seizure threshold at least 30 days prior to registration
* The patient must agree to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agree to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial and have a CD4 count >= 200 cells/microliter within 30 days prior to registration. Note: HIV testing is not required for eligibility for this protocol
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy within 30 days prior to registration, if indicated. Note: HBV viral testing is not required for eligibility for this protocol
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load within 30 days prior to registration
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Note: Any patient with a cancer (other than keratinocyte carcinoma or carcinoma in situ) who has no evidence of disease for < 3 years must contact the principal investigator, Ronald Chen, Doctor of Medicine (MD)
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry

Exclusion Criteria:

* Definitive radiologic evidence of metastatic disease (M1a, M1b or M1c) on molecular imaging (e.g. Fluciclovine F-18 PET, [FACBC, Axumin], F-18 PSMA PET [Pylarify], flotufolastat F-18 PSMA PET scan [Posluma], Gallium-68 PSMA PET scan or C-11 choline PET)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowed (completed > 3 years prior to registration)
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Androgen deprivation therapy (ADT) prior to radical prostatectomy
* Prior treatment with androgen receptor signaling inhibitor (including but not exclusive to a growing list of: abiraterone acetate, enzalutamide, apalutamide, darolutamide), unless started =< 180 days and stopped prior to registration, which is allowed
* Current use of 5-alpha reductase inhibitor. NOTE: if the alpha reductase inhibitor is stopped prior to randomization the patient is eligible
* History of any of the following:

  * Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year prior to registration, brain arteriovenous malformation, Schwannoma, meningioma, or other benign central nervous system [CNS] or meningeal disease which may require treatment with surgery or radiation therapy)
  * Severe or unstable angina, myocardial infarction, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 12 months prior to registration
  * New York Heart Association functional classification III/IV (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification.)
  * History of any condition that in the opinion of the investigator, would preclude participation in this study
* Current evidence of any of the following:

  * Known gastrointestinal disorder affecting absorption of oral medications
  * Active uncontrolled infection
  * Presence of uncontrolled hypertension (persistent systolic blood pressure [BP] >= 160 mmHg or diastolic BP >= 100 mmHg). Subjects with a history of hypertension are allowed, provided that BP is controlled to within these limits by anti-hypertensive treatment
  * Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone/prednisolone once daily
  * Baseline moderate and severe hepatic impairment (Child-Pugh Class B & C)
  * Inability to swallow oral pills
  * Any current condition that in the opinion of the investigator, would preclude participation in this study
* Patients must not plan to participate in any other therapeutic clinical trials while receiving treatment on this study
* Patients with inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival (MFS) | From randomization to detection of metastatic disease or death from any cause, assessed up to 7.5 years
  Kaplan-Meier curves will be generated and metastasis-free survival compared between the two treatment groups by a logrank test, stratified by prostate specific antigen (PSA) level after prostatectomy (never detectable or rising). Cox regression modeling to assess and adjust for the effects of PSA stratum and other baseline covariates will also be performed. The proportional hazards assumption will be tested using Schoenfeld residuals and graphical methods. Martingale residual plots will be examined to determine the best functional form for incorporating covariates into the model. A competing risks analysis will also be performed with time to distant metastasis or death from prostate cancer as the event of interest and death from other causes as the competing risk. Cumulative incidence curves will be generated along with Fine-Gray's test. Patients alive and metastasis free will be censored as of the time of the last negative examination.

SECONDARY OUTCOMES:
Quality of life (QOL) between the two treatment arms | Up to 3 years post treatment
  Quality of life scores will be derived by constructing summary measures across domains from the various quality of life instruments (Expanded Prostate Cancer Index Composite-26, EuroQol (EQ)-5 Dimension (D)-5 Level (L), Brief Pain Inventory, and Patient Reported Outcome Measurement Information System-Fatigue). Calculated health utilities will be derived from the EQ-5D-5L instrument and used to produce a quality-adjusted life year survival estimate post-treatment. The area under the curve provides an estimate of the quality-adjusted, restricted mean survival time and will be compared between the two treatment arms as described in Glasziou et al (1990). QOL scores will be analyzed using mixed effects regression for longitudinal data to compare the profiles over time between the two treatment groups (Gibbons and Hedeker, 2000). The models will include treatment, time, and treatment-by-time interaction terms as fixed effects and subjects as a random effect.
Overall survival (OS) | From randomization until date of death or censored at last date known alive, assessed up to 7.5 years
  Will be summarized by Kaplan-Meier curves and compared between treatment groups via logrank tests and Cox regression modeling.
Biochemical progression-free survival (bPFS) | From randomization until biochemical recurrence or death from prostate cancer, assessed up to 7.5 years
  Will be summarized by Kaplan-Meier curves and compared between treatment groups via logrank tests and Cox regression modeling. In addition, competing risks analyses will be performed and cumulative incidence curves generated for bPFS with death from other (i.e., non-prostate cancer) causes treated as a competing event. Patients who die from non-prostate cancer related causes will be censored as of the date of death.
Time to local-regional progression | Up to 7.5 years
  Competing risks analyses will be performed and cumulative incidence curves generated for local-regional progression with death from other (i.e., non-prostate cancer) causes treated as a competing event.
Time to castrate resistance | Up to 7.5 years
  Will be summarized by Kaplan-Meier curves and compared between treatment groups via logrank tests and Cox regression modeling. Patients who die prior to resistance will be censored.
Cancer-specific survival | Up to 7.5 years
  Will be summarized by Kaplan-Meier curves and compared between treatment groups via logrank tests and Cox regression modeling. In addition, competing risks analyses will be performed and cumulative incidence curves generated for cancer-specific survival with death from other (i.e., non-prostate cancer) causes treated as a competing event. Patients who die from non-prostate cancer related causes will be censored as of the date of death.
Incidence of adverse events | Up to 7.5 years
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0. Adverse events will be tabulated by type, level of severity, and attribution for each treatment arm and the rate of events compared between treatment groups using chi-square or Fisher's exact tests.

OTHER OUTCOMES:
MFS by Decipher genomic score | Up to 7.5 years
  Will determine the ability of the Decipher test to predict for metastasis in a purely node-positive population. Subgroup analyses of MFS by Decipher genomic score (high risk or low/intermediate risk) will be performed and tests for treatment-by-risk group interaction conducted via Cox regression to explore whether any benefits of apalutamide is limited to the high (or low/intermediate) risk stratum.
OS by Decipher genomic score | Up to 7.5 years
  Will determine the ability of the Decipher test to predict for metastasis in a purely node-positive population. Subgroup analyses of OS by Decipher genomic score (high risk or low/intermediate risk) will be performed and tests for treatment-by-risk group interaction conducted via Cox regression to explore whether any benefits of apalutamide is limited to the high (or low/intermediate) risk stratum.
PAM50-based classification of prostate cancer | Up to 7.5 years
  Will validate the PAM50-based classification of prostate cancer into luminal A, luminal B, and basal subtypes as prognostic markers. Classifications of prostate cancer into Luminal A, Luminal B, and basal subtypes using the PAM50 method of classification. Subgroup analyses will be performed and tests for treatment-by-risk group interaction conducted via Cox regression to explore whether any benefits of apalutamide is limited to the high (or low/intermediate) risk stratum.
Estimate of treatment effect by sex | Up to 7.5 years
  Estimates of the primary outcome treatment effect and the corresponding 95% confidence intervals (CIs) by sex.
Estimate of treatment effect by race | Up to 7.5 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by race.
Estimates of treatment effect by ethnicity | Up to 7.5 years
  Estimates of the primary outcome treatment effect and the corresponding 95% CIs by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald C Chen, Principal Investigator — NRG Oncology
Locations (347):
- United States (345):
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Alton Memorial Hospital, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate High Tech Medical Park, Palos Heights, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Reid Health, Richmond, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Northwell Health Physicians Partners Radiation Medicine at Queens, Forest Hills, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Garnet Health Medical Center, Middletown, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Queens Cancer Center, Rego Park, New York
  - Wilmot Cancer Institute Radiation Oncology at Greece, Rochester, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Avera Cancer Institute - Mitchell, Mitchell, South Dakota
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Tarrant County Hospital District/JPS Health Network, Fort Worth, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - VCU Massey Cancer Center at Hanover Medical Park, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (2):
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec